CLINICAL TRIAL: NCT06760416
Title: Effect of Online Diabetic Foot Support Program (DiaFootSuP) and Care Kit on Diabetic Foot Care Outcomes: Randomized Controlled Trial
Brief Title: Online Diabetic Foot Support Program- Care Kit
Acronym: DiaFootSuP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve GÃnbaAY (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Merve GÃnbaAY, Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DokuzEU-IHS-MG-01
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus; Diabetic Foot Ulcer; Diabetic Foot
Keywords: Diabetic Foot; Type 2 Diabetes; Nursing Education; Foot
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Mellitus, Type 2 | interventions — Nursing Education Research

STUDY DESIGN:
Intervention Model Description: The study is conducted by dividing patients into experimental and control groups using simple randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Groups (Experimental): 5 modules of online foot care training, motivational messages and informative videos for the patient who was given a foot care kit
  Interventions: Other: Nursing Education
- CONTROL GROUP (No Intervention): Delivery of training videos after pre-test and post-test application

INTERVENTIONS:
Other: Nursing Education — 5 modules of online foot care training, motivational messages and informative videos for the patient who was given a foot care kit
  Arms: Experimental Groups

SUMMARY:
The aim of this project is to examine the effects of the online diabetic foot support program (DiaFootSuP) and care kit applied to type 2 diabetic individuals who have previously had a diabetic foot ulcer on diabetic foot outcomes (diabetic foot knowledge level, foot care behavior level, foot care self-efficacy level, HbA1c, etc.).

DETAILED DESCRIPTION:
It was planned as a randomized controlled study to determine the effect of the online diabetic foot support program (DiaFootSuP) and care kit applied to type 2 diabetic individuals who had previously had diabetic foot ulcers on diabetic foot outcomes. The sample calculation of the study was based on determining the difference between two independent groups and the sample size for the experimental and control groups was taken as experimental: 31-control: 31 people using the G*Power 3.1.9.6 program. The experimental group was given a foot care kit developed by the researcher, which included special foot care products. Pre-test data for the experimental and control groups are collected from the diabetic foot knowledge scale, foot care behavior scale, and diabetic foot care self-efficacy scale. Online diabetic foot care training consisting of 5 modules is given individually to the patients in the experimental group. After the training, motivational messages and informative videos are sent once a week for 3 months. Patients are also asked to send photos while doing foot care. The post-test data of the experimental and control groups will be collected at the end of 3 months with the diabetic foot knowledge scale, foot care behavior scale, and diabetic foot care self-efficacy scale. Training videos will be delivered to the control group at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, Individuals diagnosed with type 2 diabetes, Patients who have had diabetic foot ulcers and have healed, Can read and write Turkish, No visual, hearing, perception and any physical disability, Physical, mental and cognitive competence to participate in self-care activities, Able to use technological products (able to use computers, tablets and smartphones), Individuals who voluntarily agree to participate in the study will constitute the sample

Exclusion Criteria:

* Patients with active diabetic foot ulcers, Individuals who cannot read or write, Individuals who cannot use technological devices, Individuals who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The 5-item Diabetes Foot Care Knowledge Scale | two week
  The 5-item Diabetes Foot Care Knowledge Scale, a subscale of the Diabetes Knowledge Questionnaire-24, was used. Cronbach's α value was found to be 0.63. Scores range from 0 to 5, with higher scores indicating higher knowledge levels.
Foot Self Care Observation Guide | two week
  The Cronbach α value of the Foot Self Care Observation Guide was determined as 0.83. The scale consists of 15 items. These items are evaluated as 1=Never, 2=Occasionally, 3=Sometimes, 4=Frequently, 5=Always. The lowest score on the scale is 15, the highest is 75. An increase in the scale score indicates that the individual's self-care behaviors are better.
Diabetic Foot Care Self Efficacy Scale | two week
  Diabetic Foot Care Self Efficacy Scale Cronbach α value was determined as 0.86. The scale consists of nine items. These nine statements are evaluated on an 11-number visual scale, which is stated as "I do not see it as sufficient at all = 0" and "I see it as very sufficient = 10". The lowest score obtained from the scale is 0, the highest score is 90. An increase in the scale score indicates that the individual has high self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Merve M GÜNBAŞ, Msc. Phd., Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No